CLINICAL TRIAL: NCT01215110
Title: A Phase II Dose Ranging Trial to Evaluate the Extended Early Bactericidal Activity, Safety, Tolerability, and Pharmacokinetics of TMC207 in Adult Patients With Newly Diagnosed, Uncomplicated, Smear-Positive, Pulmonary Tuberculosis.
Brief Title: Evaluation of Early Bactericidal Activity in Pulmonary Tuberculosis (TMC207-CL001)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Global Alliance for TB Drug Development (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TMC207-CL001
Record Dates: First submitted 2010-09-30; First posted 2010-10-06 (Estimated); Results first posted 2017-04-26 (Actual); Last update posted 2017-04-26 (Actual); Status verified 2017-01

CONDITIONS: Pulmonary Tuberculosis
Keywords: Bedaquiline; Sirturo; Early Bactericidal Activity; EBA; Pulmonary Tuberculosis; TMC207
MeSH Terms: conditions — Tuberculosis, Pulmonary | interventions — bedaquiline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- TMC207 700/500/400 (Experimental): TMC207- 700 mg Day 1; 500 mg Day 2; 400 mg Days 3-14
  Interventions: Drug: TMC207
- TMC207 500/400/300 (Experimental): TMC207- 500 mg Day 1; 400 mg Day 2 and 300 mg Days 3-14.
  Interventions: Drug: TMC207
- TMC207 400/300/200 (Experimental): TMC207- 400 mg Day 1; 300 mg Day 2 and 200 mg Days 3-14
  Interventions: Drug: TMC207
- TMC207 200/100 (Experimental): TMC207- 200 mg Day 1 and 100 mg Days 2-14
  Interventions: Drug: TMC207
- Rifafour e-275 mg (Active Comparator): Rifafour e-275 mg
  Interventions: Drug: Rifafour e-275 mg

INTERVENTIONS:
Drug: TMC207
  Arms: TMC207 200/100; TMC207 400/300/200; TMC207 500/400/300; TMC207 700/500/400
Drug: Rifafour e-275 mg
  Arms: Rifafour e-275 mg

SUMMARY:
The trial will evaluate the extended bactericidal activity of 14 consecutive days of oral administration of TMC207 at multiple doses as determined by the rate of change of log10 colony forming units (CFU) per ml sputum over the time period Day 7-14 in participants with smear positive pulmonary tuberculosis (TB). A control group will receive standard treatment.

ELIGIBILITY:
Inclusion Criteria:

* Provide written, informed consent prior to all trial-related procedures including HIV testing.
* Male or female, aged between 18 and 65 years inclusive.
* Body weight (in light clothing and with no shoes) between 40 and 90 kg, inclusive.
* Newly diagnosed, previously untreated, uncomplicated, sputum smear-positive, pulmonary TB.
* A chest X-ray picture which in the opinion of the Investigator is compatible with TB.
* Sputum positive on direct microscopy for acid-fast bacilli …(at least 1+ on the International Union Against Tuberculosis and Lung Disease (IUATLD)/World Health Organization (WHO) scale).
* Ability to produce an adequate volume of sputum as estimated from a spot assessment (estimated 10 ml or more overnight production).
* Females may participate if they are of non-childbearing potential, if they are using effective birth control methods and are willing to continue practicing birth control methods throughout treatment or if they are non-heterosexually active or willing to practice sexual abstinence throughout the treatment period or have a vasectomized partner (confirmed sterile). Therefore to be eligible for this study women of childbearing potential should either:1) use a double barrier method to prevent pregnancy (i.e. use a condom with either diaphragm or cervical cap) or 2) use hormonal based contraceptives in combination with a barrier contraceptive, or 3) use an intrauterine device in combination with a barrier contraceptive. They must also be willing to continue these contraception until 6 months after last study drug or 6 months after discontinuation from study medication in case of premature discontinuation. (Note: Hormone-based contraception may not be reliable when taking TMC207; therefore, hormone-based contraceptives cannot be used by female patients to prevent pregnancy).
* Male patients must be willing to use a condom with spermicide when having heterosexual intercourse throughout treatment and until 1 month after last study drug administration or 1 month after discontinuation from study medication in case of premature discontinuation.

Exclusion Criteria:

1. Evidence of clinically significant metabolic, gastrointestinal neurological, psychiatric or endocrine diseases, malignancy, or other abnormalities (other than the indication being studied).
2. Known or suspected hypersensitivity to study medications (including any rifamycin antibiotics)
3. Rifampicin-resistant and/or isoniazid-resistant bacteria detected with a sputum specimen collected within the pre-treatment period and tested at the study laboratory.
4. Clinically significant evidence of extrathoracic TB (miliary TB, abdominal TB, urogenital TB, osteoarthritic TB, TB meningitis), as judged by the investigator.
5. Current or past history of alcohol and/or drug use that, in the investigator's opinion, would compromise the participant's safety or compliance to the study protocol procedures.
6. HIV infected patients:

   1. having a cluster of differentiation 4 (CD4)+ count <300 cells/µL;
   2. or having received antiretroviral therapy medication within the last 90 days:
   3. or having received oral or intravenous antifungal medication within the last 90 days;
   4. or with an AIDS-defining opportunistic infection or malignancies (except pulmonary TB).
7. Significant cardiac arrhythmia requiring medication
8. Having participated in other clinical studies with investigational agents within 8 weeks prior to trial start.
9. Patients with the following QT/corrected QT(QTc) interval characteristics at screening:

   1. Marked prolongation of QT/QTc interval, e.g., confirmed demonstration of QT corrected for heart rate using Fridericia's method (QTcF) interval >450 ms at screening;
   2. History of additional risk factors for Torsade de Pointes, e.g., heart failure, hypokalemia, family history of Long QT Syndrome;
   3. Use of concomitant medications that prolong the QT/QTc interval listed as disallowed medication in Section 2.10.2;
   4. Pathological Q waves (defined as >40ms or depth >0.4-0.5mV);
   5. Evidence of ventricular pre-excitation;
   6. ECG evidence of complete or incomplete left bundle branch block or right bundle branch block;
   7. Evidence of second or third degree heart block;
   8. Intraventricular conduction delay with QRS duration >120ms;
   9. Bradycardia as defined by sinus rate <50bpm
10. Women who are pregnant or breastfeeding
11. History and/or presence (or evidence) of neuropathy or epilepsy.
12. Diabetics using insulin
13. Poor general condition where any delay in treatment cannot be tolerated per discretion of Investigator.
14. Previously received treatment with TMC207 as part of a clinical trial.
15. Treatment received with any drug active against Mycobacterium tuberculosis within 3 months prior to Visit 1.
16. Any disease or conditions in which any of the medicinal products listed in the section pertaining to prohibited medications is used.
17. Patients with the following toxicities at screening as defined by the enhanced Division of Microbiology and Infectious Disease (DMID) adult toxicity table (November 2007):

    1. creatinine grade 2 or greater (>1.5 times upper limit of normal [ULN]);
    2. lipase grade 3 or greater (>2.0 x ULN);
    3. hemoglobin grade 4 (<6.5 g/dL) except after discussion with the Medical Monitor;
    4. aspartate aminotransferase (AST) grade 4 (>8.0 x ULN) to be excluded, grade 3 (≥3.0 x ULN) must be discussed with Medical Monitor;
    5. alanine aminotransferase (ALT) grade 4 (>8.0 x ULN) to be excluded, grade 3 (≥3.0 x ULN) must be discussed with Medical Monitor;
    6. alkaline phosphatase (ALP) grade 4 (>8.0 x ULN) to be excluded, grade 3 (≥3.0 x ULN) must be discussed with Medical Monitor;
    7. total bilirubin grade 3 or greater (>2.00 x ULN, or >1.50 x ULN when accompanied by any increase in other liver function test) to be excluded, grade 2 (>1.50 x ULN, or >1.25 x ULN when accompanied by any increase in other liver function test) must be discussed with the Medical Monitor

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2010-04; Primary Completion 2010-08 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Diacon, Principal Investigator — TASK APPLIED SCIENCE, Karl Bremer Hospital
Locations (1):
- Karl Bremer Hospital, Belville, Cape Town, South Africa

RESULTS

PARTICIPANT FLOW:
Groups:
- TMC207 100: TMC207- 200 mg Day 1; and 100 mg Days 2-14
- TMC207 200: TMC207- 400 mg Day 1; 300 mg Day 2 and 200 mg Days 3-14.
- TMC207 300: TMC207- 500 mg Day 1; 400 mg Day 2 and 300 mg Days 3-14
- TMC207 400: TMC207- 700 mg Day 1; 500 mg Day 2; and 400 mg Days 3-14
- Rifafour e-275 mg: Daily Doses: 30 to 37 kg, 2 tablets; 38 to 54 kg, 3 tablets; 55 to 70 kg, 4 tablets; 71 kg and over, 5 tablets
Period: Overall Study
Arm/Group | TMC207 100 | TMC207 200 | TMC207 300 | TMC207 400 | Rifafour e-275 mg
Started | 15 | 15 | 15 | 15 | 8
Completed | 15 | 15 | 13 | 14 | 8
Not Completed | 0 | 0 | 2 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- TMC207 100: TMC207- 200 mg Day 1 and 100 mg Days 2-14
- TMC207 400: TMC207- 700 mg Day 1; 500 mg Day 2; 400 mg Days 3-14
- Total: Total of all reporting groups
Arm/Group | TMC207 100 | TMC207 200 | TMC207 300 | TMC207 400 | Rifafour e-275 mg | Total
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 8 | 68
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.5 (9.4) | 34.7 (18.1) | 31.4 (7.4) | 31.8 (10.9) | 26.1 (4.9) | 27 (11.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 7 | 5 | 2 | 24
  Male | 9 | 11 | 8 | 10 | 6 | 44
Race/Ethnicity, Customized [Number; unit: participants]
  Black | 6 | 5 | 9 | 7 | 6 | 33
  Mixed Ethnic | 9 | 10 | 6 | 8 | 2 | 35
Height [Mean (Standard Deviation); unit: meters (m)] | 1.638 (0.082) | 1.677 (0.094) | 1.674 (0.082) | 1.660 (0.057) | 1.660 (0.087) | 1.662 (0.080)
Weight at Day 1 [Mean (Standard Deviation); unit: kilograms (kg)] | 53.0 (7.74) | 52.5 (7.55) | 52.7 (8.20) | 50.6 (5.96) | 49.1 (6.69) | 51.8 (7.23)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 19.80 (2.988) | 18.63 (1.955) | 18.80 (2.754) | 18.36 (2.174) | 17.83 (2.018) | 18.77 (2.459)
HIV Status [Number; unit: participants]
  Positive | 1 | 1 | 1 | 2 | 1 | 6
  Negative | 14 | 14 | 14 | 13 | 7 | 62
Baseline log10 colony forming units (CFU) of M. Tuberculosis per ml sputum [Mean (Standard Deviation); unit: log(10) CFU/ml] | 6.302 (0.697) | 6.001 (0.903) | 6.071 (1.087) | 6.625 (0.756) | 5.995 (1.018) | 6.199 (0.892)
Baseline time to sputum culture positivity (TTP) in liquid culture media [Mean (Standard Deviation); unit: hours] | 104.8 (23.5) | 111.1 (30.6) | 115.7 (40.8) | 88.5 (10.8) | 106.7 (28.8) | 105.3 (26.9)

OUTCOME MEASURES:

1. Primary Outcome: Early Bactericidal Activity (EBA) Measured as the Mean Rate of Change of log10 Colony Forming Units (CFU) of M. Tuberculosis Per ml Sputum on Solid Medium Over Time (Days 0-14).
Description: The rates of change were calculated from the two slopes of the bi-linear (piece-wise) regression, for each treatment group. The nodes (point of inflection, i.e. where slope changes) used in these bi-linear regressions, as determined by visual inspection, were Day 3.5. node. Throughout the analyses, the established node at Day 2.5 was used in the Rifafour e-275 arm. Note that to facilitate interpretation the sign of these slopes were reversed for log10CFU/ml.
Time Frame: Fourteen consecutive days of treatment
Population: Because of insufficient data for bilinear regression, four patients were omitted from EBA(CFU) calculations.
Measure: Mean (Standard Deviation); unit: log10CFU/ml/day
Arm/Group | TMC207 100 | TMC207 200 | TMC207 300 | TMC207 400 | Rifafour e-275 mg
Number analyzed (Participants) | 14 | 15 | 13 | 14 | 8
log10CFU/ml/day | 0.040 (0.068) | 0.056 (0.051) | 0.077 (0.064) | 0.104 (0.077) | 0.112 (0.077)

2. Secondary Outcome: Early Bactericidal Activity (EBA) Measured as the Mean Rate of Change of log10 Colony Forming Units (CFU) of M. Tuberculosis Per ml Sputum on Solid Medium Over Time (Days 7-14).
Description: The rates of change were calculated from the two slopes of the bi-linear (piece-wise) regression, for each treatment group. The nodes (point of inflection, i.e. where slope changes) used in these bi-linear regressions, as determined by visual inspection, were Day 3.5. node. Throughout the analyses, the established node at Day 2.5 was used in the Rifafour e-275 arm. Since Day 7 is later than the node day, the rate of change for this outcome is equal to the slope at Day 14. Note that to facilitate interpretation the sign of these slopes were reversed for log10CFU/ml.
Time Frame: Days 7-14 of fourteen consecutive days of treatment
Population: Because of insufficient data for bilinear regression, four patients were omitted from EBA(CFU) calculations.
Measure: Mean (Standard Deviation); unit: log10CFU/ml/day
Arm/Group | TMC207 100 | TMC207 200 | TMC207 300 | TMC207 400 | Rifafour e-275 mg
Number analyzed (Participants) | 14 | 15 | 13 | 14 | 8
log10CFU/ml/day | 0.053 (0.088) | 0.086 (0.048) | 0.098 (0.084) | 0.107 (0.082) | 0.046 (0.101)

3. Secondary Outcome: Early Bactericidal Activity (EBA) Measured as the Mean Rate of Change of log10 Colony Forming Units (CFU) of M. Tuberculosis Per ml Sputum on Solid Medium Over Time (Days 2-14).
Description: as for outcome 1
Time Frame: Days 2-14 of fourteen consecutive days of treatment
Population: Because of insufficient data for bilinear regression, four patients were omitted from EBA(CFU) calculations.
Measure: Mean (Standard Deviation); unit: log10CFU/ml/day
Arm/Group | TMC207 100 | TMC207 200 | TMC207 300 | TMC207 400 | Rifafour e-275 mg
Number analyzed (Participants) | 14 | 15 | 13 | 14 | 8
log10CFU/ml/day | 0.047 (0.074) | 0.071 (0.047) | 0.088 (0.071) | 0.106 (0.078) | 0.046 (0.101)

4. Secondary Outcome: Early Bactericidal Activity (EBA) Measured as the Mean Rate of Change of log10 Colony Forming Units (CFU) of M. Tuberculosis Per ml Sputum on Solid Medium Over Time (Days 0-2).
Description: The rates of change were calculated from the two slopes of the bi-linear (piece-wise) regression, for each treatment group. The nodes (point of inflection, i.e. where slope changes) used in these bi-linear regressions, as determined by visual inspection, were Day 3.5. node. Throughout the analyses, the established node at Day 2.5 was used in the Rifafour e-275 arm. Since this range (Days0-2) is before the node day, the rate of change for this outcome is equal to the slope at Day 0. Note that to facilitate interpretation the sign of these slopes were reversed for log10CFU/ml.
Time Frame: Two consecutive days of treatment
Population: Because of insufficient data for bilinear regression, four patients were omitted from EBA(CFU) calculations.
Measure: Mean (Standard Deviation); unit: log10CFU/ml/day
Arm/Group | TMC207 100 | TMC207 200 | TMC207 300 | TMC207 400 | Rifafour e-275 mg
Number analyzed (Participants) | 14 | 15 | 13 | 14 | 8
log10CFU/ml/day | 0.004 (0.168) | -0.033 (0.128) | 0.015 (0.149) | 0.093 (0.136) | 0.413 (0.291)

5. Secondary Outcome: Rate of Change in Time to Sputum Culture Positivity (TTP)(Hours) in Liquid Culture Media (Days 0-14)
Description: The TTP was measured in the Mycobacterial Growth Indicator Tube (MGIT) (Bactec MGIT960) automated liquid culture system from overnight sputum. TTP rates of change were calculated from the two slopes of the bi-linear (piece-wise) regression, for each treatment group.
Time Frame: Fourteen consecutive days of treatment
Population: Because of insufficient data for bilinear regression, nine participants were omitted from TTP calculations.
Measure: Mean (Standard Deviation); unit: hours/day
Arm/Group | TMC207 100 | TMC207 200 | TMC207 300 | TMC207 400 | Rifafour e-275 mg
Number analyzed (Participants) | 13 | 13 | 13 | 12 | 8
hours/day | 4.0 (5.1) | 4.2 (3.1) | 4.9 (5.1) | 5.4 (3.4) | 14.3 (11.4)

6. Secondary Outcome: Rate of Change in Time to Sputum Culture Positivity (TTP)(Hours) in Liquid Culture Media (Days 0-2)
Description: as for outcome 5
Time Frame: Two consecutive days of treatment
Population: Because of insufficient data for bilinear regression, nine participants were omitted from TTP calculations.
Measure: Mean (Standard Deviation); unit: hours/day
Arm/Group | TMC207 100 | TMC207 200 | TMC207 300 | TMC207 400 | Rifafour e-275 mg
Number analyzed (Participants) | 13 | 13 | 13 | 12 | 8
hours/day | 1.5 (2.3) | 3.7 (4.3) | 4.1 (4.7) | 6.2 (3.3) | 27.3 (13.8)

7. Secondary Outcome: Rate of Change in Time to Sputum Culture Positivity (TTP)(Hours) in Liquid Culture Media (Days 2-14)
Description: as for outcome 5
Time Frame: Days 2-14 of fourteen consecutive days of treatment
Population: Because of insufficient data for bilinear regression, nine participants were omitted from TTP calculations.
Measure: Mean (Standard Deviation); unit: hours/day
Arm/Group | TMC207 100 | TMC207 200 | TMC207 300 | TMC207 400 | Rifafour e-275 mg
Number analyzed (Participants) | 13 | 13 | 13 | 12 | 8
hours/day | 4.4 (5.9) | 4.3 (3.1) | 5.1 (5.3) | 5.3 (3.5) | 11.5 (13.9)

8. Secondary Outcome: Rate of Change in Time to Sputum Culture Positivity (TTP)(Hours) in Liquid Culture Media (Days 7-14)
Description: as for outcome 5
Time Frame: Days 7-14 of fourteen consecutive days of treatment
Population: Because of insufficient data for bilinear regression, nine participants were omitted from TTP calculations.
Measure: Mean (Standard Deviation); unit: hours/day
Arm/Group | TMC207 100 | TMC207 200 | TMC207 300 | TMC207 400 | Rifafour e-275 mg
Number analyzed (Participants) | 13 | 13 | 13 | 12 | 8
hours/day | 6.9 (11.2) | 4.8 (4.4) | 5.9 (7.2) | 4.4 (5.0) | 11.5 (13.9)

9. Secondary Outcome: Summary of Statistical Analysis of TMC207 Maximum Plasma Concentration Following Dosing (C(Max)) on Days 1 and 14
Time Frame: Day 1 (0, 1, 3, 5, 6, 8, 12, and 24 hour post-dose) or Day 14 (0, 1, 3, 5, 6, 8, 12, 24, and 30 hour post-dose)
Population: On Day 14, N=13 for TMC207 300 group and N=14 for TMC207 400 group due to early withdrawal of three participants
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | TMC207 100 | TMC207 200 | TMC207 300 | TMC207 400
Number analyzed (Participants) | 15 | 15 | 15 | 15
ng/mL
  C(max) Day 1 | 1846.13 (613.55) | 2700.73 (858.54) | 3128.00 (1239.26) | 5386.67 (3069.95)
  C(max) Day 14 | 1553.27 (691.36) | 2884.67 (789.44) | 3902.31 (771.77) | 5178.57 (2663.75)

10. Secondary Outcome: Summary of Statistical Analysis of TMC207 Time of Maximum Plasma Concentration (T(Max)) on Days 1 and 14
Time Frame: Day 1 (0, 1, 3, 5, 6, 8, 12, and 24 hour post-dose) or Day 14 (0, 1, 3, 5, 6, 8, 12, 24, and 30 hour post-dose)
Population: On Day 14, N=13 for TMC207 300 group and N=14 for TMC207 400 group due to early withdrawal of three participants
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | TMC207 100 | TMC207 200 | TMC207 300 | TMC207 400
Number analyzed (Participants) | 15 | 15 | 15 | 15
hour
  T(max) Day 1 | 5.33 (1.80) | 5.20 (1.90) | 5.53 (0.83) | 5.67 (1.05)
  T(max) Day 14 | 5.13 (1.19) | 4.60 (1.06) | 5.15 (1.46) | 5.29 (1.59)

11. Secondary Outcome: Summary of Statistical Analysis of TMC207 Area Under the Concentration-time Curve Over the Dose Interval of 0 to 24 h (AUC(0-24)) on Day 1 and Day 14
Time Frame: Day 1 (0, 1, 3, 5, 6, 8, 12, and 24 hour post-dose) or Day 14 (0, 1, 3, 5, 6, 8, 12, and 24 hour post-dose)
Population: On Day 14, N=13 for TMC207 300 group and N=14 for TMC207 400 group due to early withdrawal of three participants
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | TMC207 100 | TMC207 200 | TMC207 300 | TMC207 400
Number analyzed (Participants) | 15 | 15 | 15 | 15
ng*h/mL
  AUC(0-24) Day 1 | 18995.57 (6947.92) | 26619.51 (8453.09) | 31357.35 (10596.74) | 53179.27 (20699.64)
  AUC(0-24) Day 14 | 18689.03 (4450.56) | 33314.07 (5780.02) | 50547.15 (11914.16) | 69069.64 (27062.36)

ADVERSE EVENTS:
Time Frame: 49 days
Description: Adverse events were collected by the Investigator from the time a participant signed the Informed Consent Form until the end of follow-up visit (Day 49). Data reported are treatment-emergent adverse events.
Arm/Group | TMC207 100 | TMC207 200 | TMC207 300 | TMC207 400 | Rifafour e-275 mg
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15 | 1/15 | 0/8
Other Adverse Events (participants affected / at risk) | 4/15 | 4/15 | 5/15 | 5/15 | 2/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TMC207 100 (N=15) | TMC207 200 (N=15) | TMC207 300 (N=15) | TMC207 400 (N=15) | Rifafour e-275 mg (N=8)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TMC207 100 (N=15) | TMC207 200 (N=15) | TMC207 300 (N=15) | TMC207 400 (N=15) | Rifafour e-275 mg (N=8)
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 1 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 1
Chest discomfort (General disorders) | 0 | 0 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 1
Body tinea (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 2 | 0 | 1 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 2
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator or any Sub-Investigator shall submit any oral or written publication or abstract concerning this study to the Sponsor not less than thirty (30) days prior to submission to any journal, other publication or meeting, for review and removal of confidential information.